CLINICAL TRIAL: NCT04297670
Title: Evaluation of the Impact of Quebec HPV Immunization Program: Prevalence of HPV Types in 16-20 Year Old Males
Brief Title: HPV Prevalence in 16-20 Year Old Males
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Other Study IDs: HPV2020-5037
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: HPV Infection
Keywords: Prevalence; Boys
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Self collected genital sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unvaccinated against HPV boys: Sexually active unvaccinated against HPV 16-20 years old boys.
  Interventions: Other: Measurement of HPV types prevalence

INTERVENTIONS:
Other: Measurement of HPV types prevalence — Self collected genital samples to be tested for the presence of different HPV types.

SUMMARY:
In Quebec, 18 birth cohorts of girls were vaccinated against HPV (aged 9 to 29 years in 2020). With an observed vaccination coverage of >80% an important herd effect might be expected. This study aim is to measure the HPV types prevalence in unvaccinated sexually active boys aged 16 to 20 years.

DETAILED DESCRIPTION:
An HPV immunization program is in place in Quebec since 2008. By 2020 18 birth cohorts of girls were eligible for vaccination. Vaccine uptake with at least one dose of vaccine was >80%. With such a high vaccine uptake an important herd immunity might be expected. The main objective of this study is to measure the prevalence of different HPV types in unvaccinated sexually active boys aged 16 to 20 years. This is a cross sectional study which includes one visit for all participants. Self sampling technic is used. During this phase of the study a total of 681 boys will be recruited. An additional phase of the study will be conducted at the condition that the prevalence of HPV6/11/16/18/31/33/45/52 and 58 in unvaccinated boys will be at least 8.65%. The second phase of the study if conducted will measure the prevalence of the same HPV types in 681 vaccinated boys of the same age.

ELIGIBILITY:
Inclusion Criteria:

* unvaccinated against HPV
* sexually active

Exclusion Criteria:

* received an HPV vaccine
* non sexually active

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — gender identity
Study Population: Sexually active 16-20 years old boys studying at a professional school or college.
Sampling Method: Non-Probability Sample
Enrollment: 681 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV 6/11/16/18/31/33/45/52 and 58 | Up to 18 months
  Unvaccinated sexually active 16-20 year old boys will be tested

SECONDARY OUTCOMES:
Prevalence of 31 HPV types | Up to 18 months
  Unvaccinated sexually active 16-20 year old boys will be tested

CONTACTS AND LOCATIONS:
Locations (1):
- Laval University Research Hospital Center, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any researcher outside this study

REFERENCES:
- [Derived] Wolfe C, Ionescu IG, Mayrand MH, Coutlee F, Sauvageau C. Prevalence of Human Papillomavirus Genotypes in Unvaccinated 16- to 20-Year-Old Men in Quebec, Canada. J Infect Dis. 2025 Aug 14;232(2):e203-e212. doi: 10.1093/infdis/jiaf094. PMID 39982898